CLINICAL TRIAL: NCT02686099
Title: SternaLock 360 First in Man Study: A Prospective, Randomized Controlled Trial
Brief Title: Sternal Closure With SternaLock 360: First in Man Study
Acronym: SL360
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0614
Record Dates: First submitted 2016-02-09; First posted 2016-02-19 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Sternal Fracture
Keywords: Rigid Fixation; Sternal Plating; Sternal Closure; Sternalock

STUDY DESIGN:
Intervention Model Description: Comparison of intervention using sternal closure with 360 plating system, to closure of the sternum using wire cerclage
Who Masked: Participant
Masking Description: participants are blinded to treatment choice until completion of the study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- SternaLock 360 (Experimental): Sternal closure performed with SternaLock 360 as a primary closure system
  Interventions: Device: SternaLock 360
- Wire Cerclage (Active Comparator): Sternal closure performed with standard wire cerclage as a primary closure system
  Interventions: Device: Wire Cerclage

INTERVENTIONS:
Device: SternaLock 360 — Sternal closure with SternaLock 360
  Arms: SternaLock 360
Device: Wire Cerclage — Sternal closure with standard wire cerclage
  Arms: Wire Cerclage

SUMMARY:
The SternaLock 360 Sternal Closure Device combines the techniques of rigid fixation with a cerclage material into a single sternal closure system. The cerclage material serves to facilitate sternal approximation, and the plates and screws serve to provide rigid fixation and prevent sternal movement and separation. The combination of a cerclage material in combination with plate and screw fixation may also lead to increased stability compared to either method used as a standalone means of closure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new technology for sternal closure that combines rigid plate fixation with a cerclage material in patients undergoing a cardiac surgery subsequent to a full median sternotomy. This study will evaluate intraoperative outcomes related to the surgical technique and performance of the device, sternal healing and stability, sternal wound complications and postoperative recovery (e.g. pain and functional status) in patients closed with this device. For comparative purposes, a control group of wire cerclage patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a standard midline sternotomy as a result of a cardiac surgical procedure (i.e. coronary artery bypass graft (CABG) and/or valve replacement along with other cardiac surgical procedures)
* Patients ≥ 30 years of age
* Patients who sign the Informed Consent

Exclusion Criteria: Pre-Operative

* Patients with endstage renal failure who are on dialysis or post transplant patients
* Patients taking chronic (>30 days) pre-operative narcotics
* Patients taking chronic (>30 days) steroids, immunosuppressant (including biologic immunosuppressants such as Enbrel), or chemotherapeutics (e.g. methotrexate). Patients using a steroid inhaler for asthma should not be excluded.
* Patients with confirmed HIV with a viral load of >10,000 copies
* Patients with an active infection that is currently being treated
* Patients with history or confirmed metal allergy or foreign body sensitivity
* Patients with a previous partial or full midline sternotomy
* Patients with previous radiation treatment of the chest
* Patients defined within the New York Heart Association (NYHA) or Canadian Cardiovascular Society (CCS) functional Class IV for congestive heart failure: i.e., patients with cardiac disease resulting in inability to carry on any physical activity without discomfort (CCS ; NYHA)
* Patients presenting emergent/salvage cardiac acuity as defined per the Society of Thoracic Surgeons (STS) guidelines: i.e., patients undergoing cardiopulmonary resuscitation en route to the operating room or prior to induction of anesthesia (STS)
* Patients unwilling or unable to return for follow-up

Exclusion Criteria: Operative

* Patients requiring delayed sternotomy closure
* Patients with transverse sternal fractures located beneath the cerclage band on the SternaLock 360 Device.
* Patients presenting intra-operative conditions that in the opinion of the treating surgeon would require or preclude a specific method for sternal closure, or who are not able to be closed per the protocol.
* Use of non resorbable (beeswax) bonewax along the sternotomy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-04 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Sternal Bone Healing | 6 months
  Sternal bone healing score as defined by CT scan assessment at 6 months postoperatively

SECONDARY OUTCOMES:
Sternal Pain | Baseline, postoperative day 3 to day 7, 1-month post-op, 3-month post-op and 6-month post-op
  Pain scores obtained at pre-specified time points in 4 modalities: at rest, after using incentive spirometer, after ambulation and after forced coughing. Likert scale questionnaire.
Analgesic usage | Baseline, postoperative day 0 to day 7, 1-month post-op, 3-month post-op and 6-month post-op
  Tabulation of all pain medication administered in pre-specified time points
Upper Extremities Functional Status | Baseline, 1-month post-op, 3-month post-op and 6-month post-op
  Functional status of upper extremities are evaluated using 20 items that are rated on a 5-point Likert scale known as Upper Extremity Functional Index questionnaire.
Return to Work | Baseline, 1-month post-op, 3-month post-op and 6-month post-op
  Assessment of working status of patients before and after cardiac surgery using 7-categorical question questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Hatcher, PhD, Study Director — Zimmer Biomet
Locations (1):
- Groote Schuur Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casha AR, Yang L, Kay PH, Saleh M, Cooper GJ. A biomechanical study of median sternotomy closure techniques. Eur J Cardiothorac Surg. 1999 Mar;15(3):365-9. doi: 10.1016/s1010-7940(99)00014-7. PMID 10333037
- [Background] Cohen DJ, Griffin LV. A biomechanical comparison of three sternotomy closure techniques. Ann Thorac Surg. 2002 Feb;73(2):563-8. doi: 10.1016/s0003-4975(01)03389-6. PMID 11845875
- [Background] Hirose H, Yamane K, Youdelman BA, Bogar L, Diehl JT. Rigid sternal fixation improves postoperative recovery. Open Cardiovasc Med J. 2011;5:148-52. doi: 10.2174/1874192401105010148. Epub 2011 Jul 4. PMID 21760857
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Losanoff JE, Basson MD, Gruber SA, Huff H, Hsieh FH. Single wire versus double wire loops for median sternotomy closure: experimental biomechanical study using a human cadaveric model. Ann Thorac Surg. 2007 Oct;84(4):1288-93. doi: 10.1016/j.athoracsur.2007.05.023. PMID 17888985
- [Background] Losanoff JE, Collier AD, Wagner-Mann CC, Richman BW, Huff H, Hsieh Fh, Diaz-Arias A, Jones JW. Biomechanical comparison of median sternotomy closures. Ann Thorac Surg. 2004 Jan;77(1):203-9. doi: 10.1016/s0003-4975(03)01468-1. PMID 14726062
- [Background] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Background] Pai S, Gunja NJ, Dupak EL, McMahon NL, Coburn JC, Lalikos JF, Dunn RM, Francalancia N, Pins GD, Billiar KL. A mechanical study of rigid plate configurations for sternal fixation. Ann Biomed Eng. 2007 May;35(5):808-16. doi: 10.1007/s10439-007-9272-3. Epub 2007 Mar 22. PMID 17377844
- [Background] Raman J, Lehmann S, Zehr K, De Guzman BJ, Aklog L, Garrett HE, MacMahon H, Hatcher BM, Wong MS. Sternal closure with rigid plate fixation versus wire closure: a randomized controlled multicenter trial. Ann Thorac Surg. 2012 Dec;94(6):1854-61. doi: 10.1016/j.athoracsur.2012.07.085. Epub 2012 Oct 25. PMID 23103010
- [Background] Raman J, Song DH, Bolotin G, Jeevanandam V. Sternal closure with titanium plate fixation--a paradigm shift in preventing mediastinitis. Interact Cardiovasc Thorac Surg. 2006 Aug;5(4):336-9. doi: 10.1510/icvts.2005.121863. Epub 2006 Apr 25. PMID 17670585
- [Background] Sargent LA, Seyfer AE, Hollinger J, Hinson RM, Graeber GM. The healing sternum: a comparison of osseous healing with wire versus rigid fixation. Ann Thorac Surg. 1991 Sep;52(3):490-4. doi: 10.1016/0003-4975(91)90910-i. PMID 1898136
- [Background] Schimmer C, Reents W, Berneder S, Eigel P, Sezer O, Scheld H, Sahraoui K, Gansera B, Deppert O, Rubio A, Feyrer R, Sauer C, Elert O, Leyh R. Prevention of sternal dehiscence and infection in high-risk patients: a prospective randomized multicenter trial. Ann Thorac Surg. 2008 Dec;86(6):1897-904. doi: 10.1016/j.athoracsur.2008.08.071. PMID 19022005
- [Background] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- See also: "Evaluation of Primary Plating in Sternotomy Patients for Osteosynthesis and Pain (RESTORE). — http://clinicaltrials.gov/ct2/show/study/NCT00819286?term=biomet+restore&rank=1&sect=X6015.